CLINICAL TRIAL: NCT01479270
Title: Randomized Trial of Transversus Abdominal Plane (TAP) Block at Total Laparoscopic Hysterectomy: Effect of Regional Analgesia on Quality of Recovery
Brief Title: Transversus Abdominal Plane Block at Total Laparoscopic Hysterectomy: Effect on Quality of Recovery
Acronym: TAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Robert Pollard, Clinical Fellow, Principal Investigator, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB10-01517
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Pain, Postoperative; Anesthesia
Keywords: recovery; postoperative; pain; laparoscopy; hysterectomy; ropivacaine; TAP block; local anesthesia
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP Block (Active Comparator): 20mL of 0.25% Ropivacaine with Epinephrine 1:200,000 is injected into bilateral transversus abdominal planes under ultrasound guidance.
  Interventions: Drug: TAP Block
- No Block (No Intervention): Patients randomized to this arm have band aids applied to sites on lateral abdomen without injection.

INTERVENTIONS:
Drug: TAP Block — Bilateral transversus abdominal plane injection under ultrasound guidance, done at conclusion of hysterectomy procedure, prior to emergence from general anesthesia
  Other Names: Ropivacaine with Epinephrine
  Arms: TAP Block

SUMMARY:
The Transversus Abdominal Plane (TAP) block has been used with good success to decrease postoperative pain following laparatomy. If the TAP block provides any improvement in the quality of recovery following laparoscopic hysterectomy, it could decrease the need for postoperative narcotics and allow for more outpatient hysterectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing laparoscopic hysterectomy
* Age ranges 18-80
* Reading literacy
* English speaking
* Able to give informed consent

Exclusion Criteria:

* History of relevant drug allergy
* Chronic opioid users who may have tolerance to pain medications
* Inability to understand written consent forms or give consent
* Age less than 18 or over 80
* Any conversion to open surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Kane, MD, Principal Investigator — MetroHealth Medical Center

REFERENCES:
- [Derived] Kane SM, Garcia-Tomas V, Alejandro-Rodriguez M, Astley B, Pollard RR. Randomized trial of transversus abdominis plane block at total laparoscopic hysterectomy: effect of regional analgesia on quality of recovery. Am J Obstet Gynecol. 2012 Nov;207(5):419.e1-5. doi: 10.1016/j.ajog.2012.06.052. Epub 2012 Jun 29. PMID 22840413

RESULTS

PARTICIPANT FLOW:
Groups:
- Tap Block: Patients undergoing Total Laparoscopic Hysterectomy were randomized with the Tap Block
- No Block: Patients undergoing Total Laparoscopic Hysterectomy were randomized without Tap Block
Period: Overall Study
Arm/Group | Tap Block | No Block
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tap Block; No Block: Patients randomized to either Tap Block or No Tap Block
- Total: Total of all reporting groups
Arm/Group | Tap Block | No Block | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery Questionnaire (QoR-40) on Postop Day #1 or #2
Description: 40 question survey completed on paper or by telephone on post-operative day #1 or #2, designed to measure health status after surgery and anesthesia. Scale ranges from 40 (extremely poor qualify of recovery) to 200 (excellent quality of recovery).
Time Frame: Postop Day #1 or Day #2
Measure: Median (Full Range); unit: units on a scale
Groups:
- TAP Block: 20mL of 0.25% Ropivacaine with Epinephrine 1:200,000 is injected into bilateral transversus abdominal planes under ultrasound guidance.
  TAP Block of 0.25% Ropivacaine with 1:200,000 Epinephrine: Bilateral transversus abdominal plane injection under ultrasound guidance, done at conclusion of hysterectomy procedure, prior to emergence from general anesthesia
Arm/Group | TAP Block | No Block
Number analyzed (Participants) | 28 | 28
units on a scale | 168.0 [125 to 195] | 169.5 [116 to 194]

2. Secondary Outcome: Narcotic Use
Description: narcotic use in mg of Morphine will be recorded
Time Frame: Postop Day #0 and Day #1
Measure: Median (Full Range); unit: mg of morphine
Groups:
- Tap Block; No Block: Patients undergoing Total Laparoscopic Hysterectomy were randomized to either the Tap Block or Nothing
Arm/Group | Tap Block | No Block
Number analyzed (Participants) | 28 | 28
mg of morphine
  Post operative day #0 | 11.7 [0 to 24] | 11.8 [0 to 27]
  Post operative day #1 | 7.5 [3 to 25] | 9.0 [3 to 15]

3. Secondary Outcome: Visual Analog Scale (VAS) for Pain
Description: visual analogue scales for pain will be completed on post-operative day #0 and #1, pain is assessed on a 10-point visual analogue scale (0 = no pain; 1 to 3 = mild; 4 to 6 = moderate pain; 7 to 10 = severe pain.)
Time Frame: 2 and 24 hours post operative
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tap Block | No Block
Number analyzed (Participants) | 28 | 28
units on a scale
  2 hours post operative | 5.0 [0 to 10] | 6.0 [2 to 10]
  24 hours post operative | 5.0 [0 to 8] | 5.0 [0 to 10]

4. Secondary Outcome: Intraoperative Time
Description: The total time in the operating room will be recorded to see if there is a difference between groups.
Time Frame: the total intraoperative time in minutes
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | TAP Block | No Block
Number analyzed (Participants) | 28 | 28
Minutes | 47.4 [2.4 to 108.6] | 34.5 [10.8 to 109.8]

ADVERSE EVENTS:
Arm/Group | TAP Block | No Block
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes